CLINICAL TRIAL: NCT04656353
Title: An Impact Assessment of a Culturally Tailored Online Psychosocial Self-Help Program for Chinese Immigrant Women With Breast Cancer
Brief Title: An Impact Assessment of a Culturally Tailored Online Psychosocial Program for Chinese Immigrant Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-5215.0
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chinese women; psychosocial; online program
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants randomized to the Intervention Arm will be provided with the website link to the online psychosocial program and the questionnaire and distress survey. They will be asked to use the website within two weeks and then to complete the questionnaire and distress survey after using it and mail them back in a self-addressed stamped envelope. The participants will also be asked in the 3-month follow-up questionnaire if they are interested in attending a focus group to elaborate on their experience with the psychosocial self-help program. Those who have expressed an interest will be contacted.
  Interventions: Behavioral: Intervention Arm
- Control Group (Experimental): Participants randomized to the Control group will receive standard care (no intervention). They will be used as a baseline to compare groups and assess the effect of the intervention (i.e., the online psychosocial program). At the two weeks following randomization (T1) and the 3-month follow-up periods (T2), they will be asked to complete the questionnaire and distress survey and return them in a self-addressed stamped envelope. Participants will be given two weeks to complete the questionnaire and distress survey. The same documents will be administered at the 3-month follow-up period (T2). Once the 3-month follow-up is completed, each participant will be provided with the website link to view the self-help program.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Arm — Participants randomized to the Intervention Arm will be provided with the website link to the online self-help program and a questionnaire and a distress survey. They will be asked to use the website within two weeks and then to complete these documents after using it and mail them back in a self-addressed stamped envelope. Same documents will be administered at the 3-month follow-up period, and the participant will be given two weeks to complete and return it in a self-addressed stamped envelope. Additionally, participants will also be asked in the 3-month follow-up questionnaire if they are interested in attending a focus group to elaborate on their experience with the psychosocial self-help program. Those who have expressed an interest will be contacted. The focus groups will last about 1-1.5 hours and consist of 3-4 participants. Focus groups will be audio-taped and conducted in either English or Chinese.
  Arms: Intervention Arm
Behavioral: Control Group — Participants randomized to the Control group will receive standard care (no intervention). They will be used as a baseline to compare groups and assess the effect of the intervention (i.e., the online psychosocial program). At the two weeks following randomization (T1) and the 3-month follow-up periods (T2), they will be asked to complete the questionnaire and distress survey and return them in a self-addressed stamped envelope. Participants will be given two weeks to complete the questionnaire and distress survey. The same documents will be administered at the 3-month follow-up period (T2). Once the 3-month follow-up is completed, each participant will be provided with the website link to view the self-help program.
  Arms: Control Group

SUMMARY:
The purpose of the study is to evaluate the effectiveness of an online psychosocial self-help program for Chinese immigrant women with breast cancer, by comparing Chinese immigrant women who receive the online psychosocial program and those who do not receive the program.

The investigators want to understand if this online psychosocial program is effective in helping Chinese immigrant women to feel more supported, understand that the distress is normal, engage in self-care activities, become aware of the community resources, feel more confident about returning to a normal life, and feel less distress overall as they return to life after treatment. This information will help us to better understand these Chinese immigrant women's needs and concerns and plan future growth of the program to meet their personal, cultural, and language needs.

DETAILED DESCRIPTION:
This study will be conducted over a three-year period at the Princess Margaret Cancer Centre (PM), University Health Network. The mixed-methods study design will include a longitudinal survey and a focus group component. Quantitative assessments will be conducted at three time periods: pre-intervention (T0), within 2 weeks post-intervention (T1), and three months post-intervention (T2). Two small focus groups will be conducted to deepen the understanding of the participants', who received the online psychosocial program, experience of the intervention.

The online psychosocial self-help program (www.asianbrcarecovery.ca) website is hosted with University Health Network Digital, build on the SharePoint 2013 Platform. The website is an anonymous website with open access to the general public, including Control Group participants. They may come across the online psychosocial program if they search the internet for information. A question was included in the Control Group 3-month follow-up questionnaire to track if the participants found and used the website.

Recruitment. Recruitment will be conducted by a research assistant (RA) who is fluent in English and Chinese either in-person or by telephone. The oncologist will approach each patient coming to the hospital for treatment or from virtual visits using hospital approved Ontario Telemedicine Network and introduce the study. If the participant is interested to hear more about the study, the oncologist will ask for the participant's consent to release her contact information to the RA. The RA will contact the participant and explain the nature and demands of the study, go through the informed consent form with her, and answer any questions. If the participant agrees to participate, written informed consent, Participant Demographics questionnaire, and baseline distress survey (T0) will be mailed to the participant with a return self-addressed stamped envelope prior to randomization. The two community partners (South Riverdale Community Health Center and Senior Persons Living Connected) will also help with identifying participants. The group leaders at the monthly Chinese cancer psychoeducational groups will introduce the study and if the participant is interested, they will ask for the participant's consent to have her contact information provided to the RA. The recruitment process will remain the same. The participant will be asked to complete these documents in two weeks.

Participants will be randomly assigned in a 1:1 ratio to the online psychosocial intervention (INT) or the standard care control group (CTL) by using a list of randomly generated numbers (www. Random.org): when a participant is enrolled, she will be assigned the next consecutive number in the list. Participants receiving an odd number will be assigned to the CTL condition, and those receiving an even number will be assigned to the INT condition.

Intervention Arm. Following the receipt of completed baseline (T0) questionnaires, the participants randomized to the INT group will be provided with the website link to the online psychosocial program and a questionnaire and a distress survey. They will be asked to use the website within two weeks and then complete the questionnaire and distress survey after using it (T1) and mail them back in a self-addressed stamped envelope. The RA will call participants with a reminder if completed questionnaires have not been received by the third week. The questionnaire and survey will be administered at the 3-month follow-up period (T2) either at a participant's clinic visit or by mail, and the participant will be given two weeks to complete and return it in a self-addressed stamped envelope. A reminder call will be made after the two-week period. The questionnaires will take about 10 minutes to complete.

INT participants will also be asked in the 3-month follow-up questionnaire if they are interested in attending a focus group to elaborate on their experience with the psychosocial self-help program. For those who have expressed an interest will be contacted. The focus groups will last about 1-1.5 hours and consist of 3-4 participants; the small group size will afford more focused solicitation of the primary outcomes. Focus groups will be audio-taped and conducted in either English or Chinese.

Control Group. Participants randomized to the CTL group will receive standard care. At the two weeks following randomization (T1) and the 3-month follow-up periods (T2), the RA will mail the questionnaire and distress survey for completion. Participants will be given two weeks to complete the questionnaire and distress survey. A self-addressed stamped envelope will be provided to mail them back. A reminder call will be made after the two-week period. The questionnaire and distress survey will be administered at the 3-month follow-up period (T2) either at the participant's clinic visit or by mail. The questionnaires will take about 10 minutes to complete. Once the 3-month follow-up package is received, each participant will be provided with the website link to view the self-help program.

Data Collection. Quantitative data will be collected with a pre/post measure of emotional distress (anxiety and depression), questionnaires, and website analytics (e.g., number of visits to the website per individual). All measures used in the study will be available in both English and Chinese (traditional and simplified versions), and participants will be asked about their language preference. Qualitative data will be collected from two small focus groups.

Measures. Socio-demographic and medical information will be collected with a self-report information form (Patient Demographics questionnaire) created by the research team. Any study materials that are in English (i.e., consent forms, socio-demographic information form, and questionnaires) will be professionally translated to Chinese (simplified and traditional), to accommodate the diversity in the Chinese population. The translated documents will be reviewed by the Chinese members of the team and recommendations made until acceptable Chinese-translated versions are agreed upon.

Statistical Analysis. Data will be analyzed using SPSS version 25. Participant characteristics and baseline outcome measures will be summarized using descriptive statistics. The equivalence of groups at baseline on basic demographic and medical variables will be assessed using independent t-tests and chi-square tests, and variables demonstrating any significant group differences (p<.05) will be included as covariates in the primary analyses. A data dictionary will be created containing detailed descriptions of each variable and coding information. Data checks will be verified by the study investigator.

To evaluate the effect of the online self-help program, the main and interaction effects of treatment group (INT and CTL) and time (T0, T1, and T2) on each of the primary outcomes will be examined using separate mixed ANCOVA models, controlling for any empirically identified covariates. Hedges' g and associated confidence intervals will be calculated to estimate effect sizes both over time (within groups) and between groups. Alpha will be set at 0.05, and probability values will be two-tailed. Missing data will be evaluated on a case-by-case basis such that drop-outs will be excluded.

Qualitative Data Analysis. Focus group interviews will be transcribed verbatim. Content analysis will be used to analyze focus group transcripts and identify categories and themes. Constant comparison will be undertaken by staying close to the data, identifying negative cases, and comparing themes and patterns. NVivo 10 will be used for data management.

A small honorarium will be provided to each participant at every single time period they complete the measures to compensate for the time taken to participate. Similarly, a small honorarium will be provided to the participants attending the focus groups to compensate them for their time and transportation expenses.

ELIGIBILITY:
Inclusion Criteria:

* Foreign-born Chinese immigrant women who identify their mother tongue as either Cantonese or Mandarin
* A diagnosis of new breast cancer (Stages 0-III)
* Receiving surgery (i.e., mastectomy) or adjuvant radiation therapy as the last hospital-based treatment, with the exception of Tamoxifen, bisphosphonates, and Herceptin
* Able to use a computer
* Able to read and speak English, Cantonese, or Mandarin.

Exclusion Criteria:

* recurrence or metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Changed feelings of support | Baseline, 2 weeks and 3-month periods
  A 17-item questionnaire was developed to evaluate the four primary outcomes. Each outcome variable is assessed with 4 questions that include 7-point rating scales (strongly disagree, disagree, somewhat disagree, neutral, somewhat agree, agree, and strongly agree). One multiple-choice question was included asking about the types of social/recreational activities the participant is engaged in. This questionnaire will be administered to both the Intervention Arm and Control Group. For the Intervention Arm, an additional 4 questions were included in the questionnaire at the two-week and 3-month follow-up periods asking about the impact of the online psychosocial program: the importance and usefulness of information in the website, the frequency of website visits, and the participant's interest in participating in a focus group. For the Control Group, one extra question was included in the 3-month follow-up questionnaire asking the participants if they found the website and used it.
Changed feelings of their distress as normal | Baseline, 2 weeks and 3-month periods
  A 17-item questionnaire was developed to evaluate the four primary outcomes. Each outcome variable is assessed with 4 questions that include 7-point rating scales (strongly disagree, disagree, somewhat disagree, neutral, somewhat agree, agree, and strongly agree). One multiple-choice question was included asking about the types of social/recreational activities the participant is engaged in. This questionnaire will be administered to both the Intervention Arm and Control Group. For the Intervention Arm, an additional 4 questions were included in the questionnaire at the two-week and 3-month follow-up periods asking about the impact of the online psychosocial program: the importance and usefulness of information in the website, the frequency of website visits, and the participant's interest in participating in a focus group. For the Control Group, one extra question was included in the 3-month follow-up questionnaire asking the participants if they found the website and used it.
Changed awareness of self-care activities and resources | Baseline, 2 weeks and 3-month periods
  A 17-item questionnaire was developed to evaluate the four primary outcomes. Each outcome variable is assessed with 4 questions that include 7-point rating scales (strongly disagree, disagree, somewhat disagree, neutral, somewhat agree, agree, and strongly agree). One multiple-choice question was included asking about the types of social/recreational activities the participant is engaged in. This questionnaire will be administered to both the Intervention Arm and Control Group. For the Intervention Arm, an additional 4 questions were included in the questionnaire at the two-week and 3-month follow-up periods asking about the impact of the online psychosocial program: the importance and usefulness of information in the website, the frequency of website visits, and the participant's interest in participating in a focus group. For the Control Group, one extra question was included in the 3-month follow-up questionnaire asking the participants if they found the website and used it.
Changed confidence about returning to a normal life post-treatment | Baseline, 2 weeks and 3-month periods
  A 17-item questionnaire was developed to evaluate the four primary outcomes. Each outcome variable is assessed with 4 questions that include 7-point rating scales (strongly disagree, disagree, somewhat disagree, neutral, somewhat agree, agree, and strongly agree). One multiple-choice question was included asking about the types of social/recreational activities the participant is engaged in. This questionnaire will be administered to both the Intervention Arm and Control Group. For the Intervention Arm, an additional 4 questions were included in the questionnaire at the two-week and 3-month follow-up periods asking about the impact of the online psychosocial program: the importance and usefulness of information in the website, the frequency of website visits, and the participant's interest in participating in a focus group. For the Control Group, one extra question was included in the 3-month follow-up questionnaire asking the participants if they found the website and used it.

SECONDARY OUTCOMES:
Changed emotional distress | Baseline, 2 weeks and 3month periods
  Hospital Anxiety and Depression Scale (HADS) is a 4-item scale used to assess levels of anxiety and depression in cancer populations. It is a well validated and frequently used self-reported measure consisting of a 4-point Likert rating scale ranging from 0 (not a problem) to 3 (high level of problems).

CONTACTS AND LOCATIONS:
Overall Officials: Terry Cheng, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No